CLINICAL TRIAL: NCT00224627
Title: Efficiency of Capsule Endoscopy and Push Enteroscopy in Obscure Gastrointestinal Bleeding. A Prospective Randomized Study.
Brief Title: Capsule Endoscopy vs. Push Enteroscopy in Occult Gastrointestinal Bleeding OGIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P040101; CDT03002
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Occult Gastrointestinal Bleeding
Keywords: Randomized study; Capsule endoscopy; Push enteroscopy; Occult gastrointestinal bleeding; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Capsule GIVEN IMAGING LTD

SUMMARY:
Capsule endoscopy (CE) is a safe and effective tool for the assessment of obscure gastrointestinal bleeding (OGIB). However, its real efficacy and its position in the diagnostic algorithm of OGIB vs. push enteroscopy (PE) remain unknown since in previous studies both techniques were performed in all included patients The purpose of this protocol is to conduct a randomized prospective controlled trial in patients with OGIB comparing a strategy based on CE or PE followed by the alternative exploration only when the first line exploration was negative. The main outpoint of this study concerns the diagnostic yield of the two explorations. Second endpoint concerns the clinical relevance of the two strategies tested (CE ± PE vs. CE ± PE) in terms of diagnostic yield, clinical outcome, therapeutic impact and added explorations

DETAILED DESCRIPTION:
This was a prospective randomized multicentric study. After the screening visit, eligible subjects were randomly assigned to be explored by CE or PE (first line exploration). The alternative exploration was only performed if no diagnosis was evidenced by the examination assigned by randomization. An independent staff member assigned subjects in 1:1 ratio between CE and PE strategies with stratification for overt and occult bleeding and centers according to consecutive number that were kept in serialized sealed opaque envelopes. After the completion of these explorations, the patients returned at month 3, 6 and 12 thereafter. At each visit, clinical evaluation and laboratory tests were performed and patients were managed according to published recommendations2 (AGA medical position). The first line exploration as well as the alternative exploration could be done during the one year follow-up period only in case of severe relapse of OGIB or necessity to perform biopsies or a therapeutic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients may suffer from episodes of active bleeding within the last 6 months or chronic iron-deficiency anemia (hemoglobin < 10 g/dl).
* A gynecologic or proctologic bleeding source had to be excluded.
* All patients had to have negative workup including upper gastrointestinal endoscopy, colonoscopy and small-bowel barium series or computed tomography enteroclysis.
* Medical reports and/or the imaging documents were available and reviewed in all patients. Usually these investigations were repeated several times before inclusion.
* Abdominal angiography was only performed when there were signs of active bleeding during the diagnostic work-up (n = 3). Meckel scintigraphy was usually carried out in patients under 30 years of age (n = 14).

Exclusion Criteria:

* Patient presenting a digestive bleeding with an echo hemodynamic major and\or requiring urgent therapeutic measures
* Wait presenting a gynaecological cause or a cause proctology of sure imputability or syndrome of malabsorption or deficiency of contribution not formally excluded
* Patient presenting an occlusive syndrome or a hurt of stenosis hail objectivized by a radiological exploration
* Surrounding wall(Speaker) or in age waits to procreate without effective contraception
* The mental or physical state of the patient not allowing a maid compliance in the conditions of the try(essay) and or in the correct use of the device Patient carrier of a pacemaker or another electromechanical implant
* Patient that must undergo an examination by MRI before having been able to eliminate the capsule
* Enteroscopy or video capsule prerequisite technically satisfactory and in touch with same pathological episode or dating at least less than 6 months Patient participating at present in another clinical trial without direct profit which can directly or indirectly influence the results(profits) of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2002-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary end point was the diagnostic yield of CE and PE (first line exploration allocated by randomization) for the identification of a definitive source of bleeding.

SECONDARY OUTCOMES:
Secondary end points were evaluated at the end of the follow up period and concerned the clinical relevance of the two strategies (PE ± CE vs. CE ± PE). They included: (1) the diagnostic yield of the two strategies for the identification of a definitive

CONTACTS AND LOCATIONS:
Overall Officials: Raymond JIAN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Adler DG, Knipschield M, Gostout C. A prospective comparison of capsule endoscopy and push enteroscopy in patients with GI bleeding of obscure origin. Gastrointest Endosc. 2004 Apr;59(4):492-8. doi: 10.1016/s0016-5107(03)02862-1. PMID 15044884